CLINICAL TRIAL: NCT03014479
Title: Study of the QOL Evaluation of Trelagliptin in Patients With Type 2 Diabetes Mellitus
Acronym: TRENDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trelagliptin-4002; JapicCTI-173482 (Registry Identifier: JapicCTI); U1111-1189-9256 (Registry Identifier: WHO)
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trelagliptin (Experimental): Trelagliptin 100 mg, orally, once weekly for up to 12 weeks. Trelagliptin 50 mg, orally, once weekly for up to 12 weeks in patients with moderate renal impairment.
  Interventions: Drug: Trelagliptin
- Daily DPP-4 inhibitors (Active Comparator): An inhibitor orally administered at the dosage and administration in the package inserts for each drug, for up to 12 weeks.
  Interventions: Drug: Daily DPP-4 inhibitor

INTERVENTIONS:
Drug: Trelagliptin — Trelagliptin 100 mg or 50 mg
  Arms: Trelagliptin
Drug: Daily DPP-4 inhibitor — Alogliptin, anagliptin, linagliptin, saxagliptin, sitagliptin, teneligliptin or vildagliptin
  Arms: Daily DPP-4 inhibitors

SUMMARY:
The purpose of this study is to assess the reduction in treatment burden during 12 weeks of trelagliptin administration in patients with type 2 diabetes on diet and exercise therapy only.

DETAILED DESCRIPTION:
The purpose of this study is to assess the reduction in treatment burden during 12 weeks of trelagliptin administration in patients with type 2 diabetes on diet and exercise therapy only. Eligible participants will be randomized to either the study drug (trelagliptin) group or the comparative drug (daily DPP-4 inhibitor) group. Treatment burden will be assessed using Diabetes Therapy Related -QOL (DTR-QOL) questionnaire and Diabetes Treatment Satisfaction Questionnaire (DTSQ).

ELIGIBILITY:
Inclusion Criteria:

1. Participants diagnosed as type 2 diabetes.
2. Participants with a stable diet and exercise therapy only for at least 12 weeks prior to the start of the screening period.
3. Participants who require a DPP-4 inhibitor treatment.
4. Participants with Hemoglobin A1c (HbA1c) >=6.5 % and <10.0 % at the start of the screening period.
5. Participants who completed DTR-QOL questionnaire at the start of the screening period.
6. Participants who have received less than 2 types of medication for treatment of comorbidities (such as hypertension or dyslipidemia) at the start of the screening period (any number of daily doses).
7. Participants who, in the opinion of the principal investigator or the investigator, are capable of understanding the content of the clinical study and complying with the study protocol requirements.
8. Participants who can provide the written informed consent prior to the initiation of any study procedures.
9. Participants aged >=20 years at the time of informed consent.
10. Outpatient.

Exclusion Criteria:

1. Participants who are receiving any oral anti-diabetic medication for the treatment of type 2 diabetes at the start of the screening period.
2. Participants diagnosed with type 1 diabetes.
3. Participants with severe renal impairment or renal failure (e.g., estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m^2 or on dialysis).
4. Participants with serious heart disease or cerebrovascular disorder, or serious pancreatic, blood, or other disease.
5. Participants with a history of gastrointestinal resection.
6. Participant with a proliferative diabetic retinopathy.
7. Participant with malignancy.
8. Participants with a history of hypersensitivity or allergy to DPP-4 inhibitors.
9. Pregnant, lactating or planning pregnancy during the study period.
10. Participants who may need to add or discontinue concomitant medication or change the dose during the study period.
11. Participants who will require treatment with a prohibited concomitant medication during the study period.
12. Participants participating in other clinical studies.
13. Participants assessed ineligible in the study by the principal investigator or the investigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2017-02-18 (Actual); Primary Completion 2017-10-21 (Actual); Study Completion 2017-10-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (27):
- Japan (27):
  - Takeda Selected Site 17, Nagoya, Aichi-ken
  - Takeda Selected Site 18, Nagoya, Aichi-ken
  - Takeda Selected Site 25, Obata, Gunma
  - Takeda Selected Site 9, Kobe, Hyōgo
  - Takeda Selected Site 27, Koga, Ibaraki
  - Takeda Selected Site 14, Kawasaki, Kanagawa
  - Takeda Selected Site 11, Sagamihara, Kanagawa
  - Takeda Selected Site 10, Yamato, Kanagawa
  - Takeda Selected Site 4, Sendai, Miyagi
  - Takeda Selected Site 5, Sendai, Miyagi
  - Takeda Selected Site 3, Kashihara, Nara
  - Takeda Selected Site 15, Kashihara, Osaka
  - Takeda Selected Site 1, Suita, Osaka
  - Takeda Selected Site 24, Okegawa, Saitama
  - Takeda Selected Site 26, Oyama, Tochigi
  - Takeda Selected Site 23, Adachi-ku, Tokyo
  - Takeda Selected Site 6, Chuo-ku, Tokyo
  - Takeda Selected Site 7, Chuo-ku, Tokyo
  - Takeda Selected Site 22, Edogawa-ku, Tokyo
  - Takeda Selected Site 19, Musashino, Tokyo
  - Takeda Selected Site 21, Ōta-ku, Tokyo
  - Takeda Selected Site 12, Shibuya-ku, Tokyo
  - Takeda Selected Site 13, Shinagawa-ku, Tokyo
  - Takeda Selected Site 20, Shinagawa-ku, Tokyo
  - Takeda Selected Site 2, Shinjuku-ku, Tokyo
  - Takeda Selected Site 8, Shinjuku-ku, Tokyo
  - Takeda Selected Site 16, Osaka

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Ishii H, Suzaki Y, Miyata Y, Matsui S. Randomized Multicenter Evaluation of Quality of Life and Treatment Satisfaction in Type 2 Diabetes Patients Receiving Once-Weekly Trelagliptin Versus a Daily Dipeptidyl Peptidase-4 Inhibitor. Diabetes Ther. 2019 Aug;10(4):1369-1380. doi: 10.1007/s13300-019-0643-1. Epub 2019 Jun 18. PMID 31214997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in Japan, from 18 February 2017 to 21 October 2017.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus on diet and exercise therapy only, were enrolled in 1 of 2 treatment groups (Trelagliptin once-weekly, or the Daily DPP-4 inhibitor once- or twice-daily (according to individual label instructions), orally, for up to 12 weeks).
Period: Overall Study
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Started | 110 | 109
Completed | 110 | 105
Not Completed | 0 | 4
Not completed — Adverse Event | 0 | 1
Not completed — Voluntary Withdrawal | 0 | 2
Not completed — Unacceptable Inability of Site Visit | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): All participants who were randomized and received at least 1 dose of the study drug for the treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors | Total
Number analyzed (Participants) | 110 | 108 | 218
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (8.96) | 58.4 (10.01) | 59.9 (9.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 26 | 50
  Male | 86 | 82 | 168
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: Participants]
  Japan | 110 | 108 | 218
Height [Mean (Standard Deviation); unit: Centimeter (cm)] | 165.0 (9.56) | 165.6 (9.29) | 165.3 (9.41)
Weight [Mean (Standard Deviation); unit: Kilogram (kg)] | 67.57 (11.917) | 70.51 (15.707) | 69.03 (13.969)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter (kg/m^2)] — Body Mass Index = weight (kg)/[height (m)^2]
  Kilogram per square meter (kg/m^2) | 24.72 (3.224) | 25.53 (4.349) | 25.12 (3.836)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 48 | 40 | 88
  Current smoker | 24 | 28 | 52
  Ex-smoker | 38 | 40 | 78
Alcohol Classification [Count of Participants; unit: Participants] — Participants who answered Yes or No for a question "Drink Alcohol Almost Every Day?" were reported.
  Participants
    Yes | 38 | 36 | 74
    No | 72 | 72 | 144
Duration of type 2 diabetes mellitus [Mean (Standard Deviation); unit: Years] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  Years | 6.45 (4.972) | 6.39 (5.286) | 6.42 (5.118)
Any Medication for Concurrent Condition [Count of Participants; unit: Participants] — Number of participants who received any medication for concurrent condition was reported.
  Participants
    Had Any Medication | 50 | 41 | 91
    Had No Any Medication | 60 | 67 | 127
Number of Daily Doses of Medication (Concurrent Condition Medicine.) [Count of Participants; unit: Participants] — Population: The baseline characteristic was analyzed in participants who had any medication for concurrent condition.
  Participants
    number analyzed (Participants) | 50 | 41 | 91
    Less than (<) 2 Times | 46 | 39 | 85
    Greater than or Equal to (≥) 2 Times | 4 | 2 | 6
Total Number of Daily Tablets (Concurrent Condition Medicine.) [Count of Participants; unit: Participants] — Population: The baseline characteristic was analyzed in participants who had any medication for concurrent condition.
  Participants
    number analyzed (Participants) | 50 | 41 | 91
    <2 Tablets | 44 | 38 | 82
    ≥2 Tablets | 6 | 3 | 9
Number of Doses of Drugs (Study drug.) [Count of Participants; unit: Participants]
  Once a Week | 110 | 0 | 110
  Once daily | 0 | 100 | 100
  Twice daily | 0 | 8 | 8
Glycated hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 7.37 (0.730) | 7.37 (0.624) | 7.37 (0.678)
DTR-QOL Total Score at Week-4 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 66.41 (15.934) | 66.37 (14.725) | 66.39 (15.311)
DTR-QOL Total Score at Week 0 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 68.48 (17.158) | 68.86 (16.240) | 68.67 (16.673)
DTR-QOL Total Score; Factor 1 at Week 0 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 73.31 (20.934) | 73.48 (20.060) | 73.39 (20.459)
DTR-QOL Total Score; Factor 2 at Week 0 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 62.94 (20.334) | 65.10 (19.725) | 64.01 (20.018)
DTR-QOL Total Score; Factor 3 at Week 0 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 79.13 (24.721) | 78.97 (23.254) | 79.05 (23.950)
DTR-QOL Total Score; Factor 4 at Week 0 [Mean (Standard Deviation); unit: Units on a Scale] — DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL including 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13; number of questions), Factor 2: Anxiety and dissatisfaction with treatment (8), Factor 3: Hypoglycemia (4) and Factor 4: Treatment satisfaction (4). Each item is scored ranging from 1 to 7 and will be added up, and summed scores will be converted from 0 (worst) to 100 (best). Higher scores reflect better QOL and positive changes from baseline indicate improvement of QOL.
  Units on a Scale | 53.22 (16.539) | 51.27 (16.347) | 52.26 (16.435)
DTSQ Total score [Mean (Standard Deviation); unit: Units on a Scale] — The DTSQ is a self-reported instrument consists of 6 questions about treatment satisfaction and 2 questions regarding blood sugar level. Each question answered on a 7-point Likert scale from 0 to 6, based on concern with the diabetes treatment and experiences in the past few weeks. Higher total score for questions about treatment satisfaction indicate greater satisfaction with treatment and experiences. Population: The number analyzed is the number of participants with data available for analysis.
  Units on a Scale
    number analyzed (Participants) | 108 | 108 | 216
    (all) | 22.31 (5.444) | 21.56 (5.679) | 21.94 (5.562)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Score for All Question Items in the Diabetes Therapy Related -QOL (DTR-QOL) Questionnaire at the End of Study
Description: DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL. It includes 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13 questions), Factor 2: Anxiety and dissatisfaction with treatment (8 questions), Factor 3: Hypoglycemia (4 questions) and Factor 4: Treatment satisfaction (4 questions). Each item is scored ranging from 1 to 7. Every score of the questions in Factor 1-3 and the score in Factor 4 converted into reverse (1-7 will be converted to 7-1) will be simply added up, and scores of each factor and the total figure will be subsequently converted from 0 to 100 (the best and worst scores will be equivalent to 100 and 0). Higher scores reflect better QOL and positive changes relative to baseline indicate improvement of QOL.
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale | 8.72 (16.162) | 6.35 (14.093)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.2305, ANCOVA; Differences of Least Square Means = 2.418, 95% CI 2-sided [-1.546 to 6.382] — Trelagliptin - Daily DPP-4 inhibitors

2. Secondary Outcome: Change From Baseline in Total Score for Each Factor Provided Through the DTR-QOL Questionnaire [Factor 1: Burden on Social Activities and Daily Activities] at Each Assessment Time Point
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to Week 4, 12, and the end of study (Week 12)
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. The number analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | 11.24 (18.200) | 7.83 (19.426)
  Week 12: number analyzed (Participants) | 109 | 105
  Week 12 | 10.98 (20.116) | 9.12 (18.560)
  End of Study | 10.79 (20.126) | 8.92 (19.048)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.4536, ANCOVA; Differences of Least Square Means = 1.938, 95% CI 2-sided [-3.150 to 7.027] — Trelagliptin - Daily DPP-4 inhibitors

3. Secondary Outcome: Change From Baseline in Total Score for Each Factor Provided Through the DTR-QOL Questionnaire [Factor 2: Anxiety and Dissatisfaction With Treatments] at Each Assessment Time Point
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to Week 4, 12, and the end of study (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | 5.18 (14.925) | 0.39 (13.769)
  Week 12: number analyzed (Participants) | 109 | 105
  Week 12 | 5.94 (18.577) | 2.18 (17.498)
  End of Study | 6.23 (18.735) | 2.10 (17.315)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.0896, ANCOVA; Differences of Least Square Means = 4.160, 95% CI 2-sided [-0.649 to 8.968] — Trelagliptin - Daily DPP-4 inhibitors

4. Secondary Outcome: Change From Baseline in Total Score for Each Factor Provided Through the DTR-QOL Questionnaire [Factor 3: Hypoglycemia] at Each Assessment Time Point
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to Week 4, 12, and the end of study (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | 6.15 (23.155) | 4.87 (22.298)
  Week 12: number analyzed (Participants) | 109 | 105
  Week 12 | 5.85 (22.837) | 7.38 (21.224)
  End of Study | 6.06 (22.840) | 6.67 (21.586)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.8506, ANCOVA; Differences of Least Square Means = -0.563, 95% CI 2-sided [-6.448 to 5.323] — Trelagliptin - Daily DPP-4 inhibitors

5. Secondary Outcome: Change From Baseline in Total Score for Each Factor Provided Through the DTR-QOL Questionnaire [Factor 4: Satisfaction With Treatment] at Each Assessment Time Point
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to Week 4, 12, and the end of study (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | 5.24 (22.254) | 3.85 (17.143)
  Week 12: number analyzed (Participants) | 108 | 105
  Week 12 | 8.53 (23.607) | 6.71 (18.431)
  End of Study | 8.86 (23.806) | 6.17 (18.507)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.3533, ANCOVA; Differences of Least Square Means = 2.696, 95% CI 2-sided [-3.018 to 8.410] — Trelagliptin - Daily DPP-4 inhibitors

6. Secondary Outcome: Change From Baseline in Total Score for All Question Items in the DTR-QOL Questionnaire at Each Assessment Time Point
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to Week 4, 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 109 | 106
  Week 4 | 8.04 (13.111) | 4.82 (12.776)
  Week 12: number analyzed (Participants) | 108 | 105
  Week 12 | 8.58 (16.280) | 6.63 (14.046)

7. Secondary Outcome: Change From Baseline in Total Score for Questions About Treatment Satisfaction in the Diabetes Treatment Satisfaction Questionnaire (DTSQ) at Each Assessment Time Point
Description: The DTSQ is a self-reported instrument consists of 6 questions about treatment satisfaction and 2 questions regarding blood sugar level. Each question answered on a 7-point Likert scale from 0 to 6, based on concern with the diabetes treatment and experiences in the past few weeks. Higher total score for questions about treatment satisfaction indicate greater satisfaction with treatment and experiences.
Time Frame: Baseline (Week 0), up to Week 4, 12 and the end of study (Week 12)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Week 4: number analyzed (Participants) | 108 | 106
  Week 4 | 3.1 (6.35) | 1.7 (6.15)
  Week 12: number analyzed (Participants) | 107 | 105
  Week 12 | 3.1 (7.59) | 2.9 (6.88)
  End of Study: number analyzed (Participants) | 108 | 108
  End of Study | 3.1 (7.59) | 2.5 (7.20)
Statistical Analysis 1: Comparison: Trelagliptin vs Daily DPP-4 Inhibitors; Test type: Superiority; p = 0.5451, ANCOVA; Differences of Least Square Means = 0.613, 95% CI 2-sided [-1.380 to 2.605] — Trelagliptin - Daily DPP-4 inhibitors

8. Secondary Outcome: Change From Baseline in Total Score for All Question Items in the DTR-QOL Questionnaire at the End of Study Stratified by the Use of Medication for Treatment of Comorbidities at Baseline
Description: DTR-QOL Questionnaire is a self-reported instrument assessing impact of diabetes treatment on health-related QOL. It includes 29 items across 4 subscales; Factor 1: Burden on social activities and daily activities (13 questions), Factor 2: Anxiety and dissatisfaction with treatment (8 questions), Factor 3: Hypoglycemia (4 questions) and Factor 4: Treatment satisfaction (4 questions). Each item is scored ranging from 1 to 7. Every score of the questions in Factor 1-3 and the score in Factor 4 converted into reverse (1-7 will be converted to 7-1) will be simply added up, and scores of each factor and the total figure will be subsequently converted from 0 to 100 (the best and worst scores will be equivalent to 100 and 0). Higher scores reflect better QOL and positive changes relative to baseline indicate improvement of QOL. Reported data was the score stratified by the use of medication for treatment of comorbidities at baseline (Used/ Not used).
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Used: number analyzed (Participants) | 50 | 41
  Used | 6.46 (15.728) | 5.80 (11.364)
  Not used: number analyzed (Participants) | 60 | 67
  Not used | 10.60 (16.408) | 6.68 (15.603)

9. Secondary Outcome: Change From Baseline in Total Score for Questions About Treatment Satisfaction in the DTSQ at the End of Study Stratified by the Use of Medication for Treatment of Comorbidities at Baseline
Description: The DTSQ is a self-reported instrument consists of 6 questions about treatment satisfaction and 2 questions regarding blood sugar level. Each question answered on a 7-point Likert scale from 0 to 6, based on concern with the diabetes treatment and experiences in the past few weeks. Higher total score for questions about treatment satisfaction indicate greater satisfaction with treatment and experiences. Reported data was the score stratified by the use of medication for treatment of comorbidities at baseline (Used/ Not used).
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. The number analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 108 | 108
Units on a Scale
  Used: number analyzed (Participants) | 50 | 41
  Used | 1.7 (8.44) | 1.2 (4.52)
  Not used: number analyzed (Participants) | 58 | 67
  Not used | 4.3 (6.61) | 3.3 (8.37)

10. Secondary Outcome: Change From Baseline in Total Score for All Question Items in the DTR-QOL Questionnaire at the End of Study Stratified by the Number of Daily Doses of Medication for Treatment of Comorbidities (<2 Times or ≥2 Times) at Baseline
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. This outcome measure was analyzed with FAS in participants who had any medication for concurrent condition at baseline.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 50 | 41
Units on a Scale
  <2 times: number analyzed (Participants) | 46 | 39
  <2 times | 6.26 (16.035) | 5.57 (11.519)
  ≥2 times: number analyzed (Participants) | 4 | 2
  ≥2 times | 8.76 (13.259) | 10.34 (8.940)

11. Secondary Outcome: Change From Baseline in Total Score for Questions About Treatment Satisfaction in the DTSQ at the End of Study Stratified by the Number of Daily Doses of Medication for Treatment of Comorbidities (<2 Times or ≥2 Times) at Baseline
Description: as for outcome 7
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 50 | 41
Units on a Scale
  <2 times: number analyzed (Participants) | 46 | 39
  <2 times | 1.3 (8.29) | 1.2 (4.58)
  ≥2 times: number analyzed (Participants) | 4 | 2
  ≥2 times | 6.8 (9.71) | 2.0 (4.24)

12. Secondary Outcome: Change From Baseline in Total Score for All Question Items in the DTR-QOL Questionnaire at the End of Study Stratified by the Total Number of Daily Tablets of Medication for Treatment of Comorbidities (<2 Tablets or ≥2 Tablets) at Baseline
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 50 | 41
Units on a Scale
  <2 tablets: number analyzed (Participants) | 44 | 38
  <2 tablets | 5.72 (16.048) | 6.00 (11.346)
  ≥2 tablets: number analyzed (Participants) | 6 | 3
  ≥2 tablets | 11.88 (13.008) | 3.26 (13.809)

13. Secondary Outcome: Change From Baseline in Total Score for Questions About Treatment Satisfaction in the DTSQ at the End of Study Stratified by the Total Number of Daily Tablets of Medication for Treatment of Comorbidities (<2 Tablets or ≥2 Tablets) at Baseline
Description: as for outcome 7
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 50 | 41
Units on a Scale
  <2 tablets: number analyzed (Participants) | 44 | 38
  <2 tablets | 1.1 (8.42) | 1.2 (4.64)
  ≥2 tablets: number analyzed (Participants) | 6 | 3
  ≥2 tablets | 6.3 (7.71) | 1.7 (3.06)

14. Secondary Outcome: Change From Baseline in Total Score for All Question Items in the DTR-QOL Questionnaire at the End of Study Stratified by the Number of Doses of the Study Drug or Comparative Drug (Once Weekly, Once Daily or Twice Daily) at Baseline
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: Full analysis set (FAS); FAS was defined as participants who were randomized and received at least one dose of the study drug. The number analyzed is the number of participants with data available for analysis at the given population.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Once Weekly: number analyzed (Participants) | 110 | 0
  Once Weekly | 8.72 (16.162) |
  Once Daily: number analyzed (Participants) | 0 | 100
  Once Daily |  | 6.90 (14.204)
  Twice Daily: number analyzed (Participants) | 0 | 8
  Twice Daily |  | -0.50 (11.176)

15. Secondary Outcome: Change From Baseline in Total Score for Questions About Treatment Satisfaction in the DTSQ at the End of Study Stratified by the Number of Doses of the Study Drug or Comparative Drug (Once Weekly, Once Daily or Twice Daily) at Baseline
Description: as for outcome 7
Time Frame: Baseline (Week 0), up to the end of study (Week 12)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 108 | 108
Units on a Scale
  Once Weekly: number analyzed (Participants) | 108 | 0
  Once Weekly | 3.1 (7.59) |
  Once Daily: number analyzed (Participants) | 0 | 100
  Once Daily |  | 2.8 (6.73)
  Twice Daily: number analyzed (Participants) | 0 | 8
  Twice Daily |  | -0.5 (11.89)

16. Secondary Outcome: Change From Baseline in Score Per Question in the DTR-QOL Questionnaire at the End of Study
Description: as for outcome 1
Time Frame: Baseline (Week 0), up to end of study (Week 12)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Units on a Scale
  Question Number 1 | 0.9 (2.39) | 0.5 (1.89)
  Question Number 2 | 1.0 (2.25) | 0.7 (1.73)
  Question Number 3 | 0.5 (1.89) | 0.2 (1.76)
  Question Number 4 | 0.7 (2.27) | 0.5 (1.72)
  Question Number 5 | 0.3 (1.73) | 0.4 (1.42)
  Question Number 6 | 0.6 (1.90) | 0.5 (1.80)
  Question Number 7 | 0.9 (1.83) | 0.7 (1.88)
  Question Number 8 | 0.8 (1.80) | 1.0 (1.75)
  Question Number 9 | 0.8 (1.85) | 0.5 (1.97)
  Question Number 10 | 0.7 (1.64) | 0.5 (1.52)
  Question Number 11 | 0.3 (1.71) | 0.3 (1.59)
  Question Number 12 | 0.6 (1.54) | 0.5 (1.29)
  Question Number 13 | 0.5 (1.59) | 0.6 (1.42)
  Question Number 14 | 0.5 (1.62) | 0.4 (1.75)
  Question Number 15 | 0.3 (1.75) | 0.3 (1.69)
  Question Number 16 | 0.4 (1.54) | 0.5 (1.31)
  Question Number 17 | 0.3 (1.44) | 0.4 (1.42)
  Question Number 18 | 0.5 (1.65) | 0.4 (1.47)
  Question Number 19 | 0.2 (1.72) | 0.2 (1.35)
  Question Number 20 | 0.5 (1.95) | 0.1 (1.93)
  Question Number 21 | 0.4 (1.72) | 0.0 (1.62)
  Question Number 22 | 0.6 (1.71) | 0.1 (1.92)
  Question Number 23 | 0.4 (1.81) | 0.1 (1.60)
  Question Number 24 | 0.2 (1.91) | 0.1 (1.65)
  Question Number 25 | 0.2 (1.68) | 0.0 (1.43)
  Question Number 26 | 0.7 (1.89) | 0.4 (1.49)
  Question Number 27 | 0.4 (1.77) | 0.3 (1.48)
  Question Number 28 | 0.3 (1.69) | 0.3 (1.33)
  Question Number 29 | 0.8 (1.59) | 0.4 (1.40)

17. Secondary Outcome: Change From Baseline in Score Per Question in the the DTSQ at the End of Study
Description: as for outcome 7
Time Frame: Baseline (Week 0), up to end of study (Week 12)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 108 | 108
Units on a Scale
  Question Number 1 | 0.7 (1.50) | 0.6 (1.47)
  Question Number 2 | -0.4 (1.77) | -0.5 (2.08)
  Question Number 3 | 0.0 (1.54) | -0.2 (1.76)
  Question Number 4 | 0.8 (1.57) | 0.5 (1.60)
  Question Number 5 | 0.6 (1.61) | 0.5 (1.47)
  Question Number 6 | 0.1 (1.47) | 0.2 (1.39)
  Question Number 7 | 0.5 (1.51) | 0.3 (1.25)
  Question Number 8 | 0.5 (1.44) | 0.4 (1.56)

18. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Participants | 19 | 20

19. Secondary Outcome: Number of Participants Reporting One or More Hypoglycemia
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Participants | 0 | 0

20. Secondary Outcome: Duration of Hospitalization for Type 2 Diabetes (Excluding Educational Hospitalization Without Worsening of Diabetes)
Description: The investigators checked any hospitalization of study participants for type 2 diabetes after the first administration of the study drug or comparative drug (excluding educational hospitalization without worsening of diabetes).
Time Frame: Up to 12 weeks
Population: There were no participants with hospitalization related to type 2 diabetes mellitus during this study.
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: Number of Participants With Hospitalization for Type 2 Diabetes (Excluding Educational Hospitalization Without Worsening of Diabetes)
Time Frame: Up to 12 weeks
Population: Safety Analysis Set: All participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
Number analyzed (Participants) | 110 | 108
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 12
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Trelagliptin | Daily DPP-4 Inhibitors
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/108
Serious Adverse Events (participants affected / at risk) | 2/110 | 0/108
Other Adverse Events (participants affected / at risk) | 4/110 | 2/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin (N=110) | Daily DPP-4 Inhibitors (N=108)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trelagliptin (N=110) | Daily DPP-4 Inhibitors (N=108)
Viral upper respiratory tract infection (Infections and infestations) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-07-05): https://cdn.clinicaltrials.gov/large-docs/79/NCT03014479/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03014479/SAP_001.pdf